CLINICAL TRIAL: NCT04415749
Title: A Double-blind, Randomized, Placebo-controlled, Study of the Safety and Immunogenicity of NasoShield Administered as One or Two Doses in Different Dosing Positions
Brief Title: NasoShield in Healthy Adults to Study Safety and Immunogenicity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Altimmune, Inc. (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ALT-201-102; HHSO100201600008C (Other Grant/Funding Number: BARDA)
Record Dates: First submitted 2020-06-01; First posted 2020-06-04 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Healthy Volunteers
Keywords: Anthrax
MeSH Terms: conditions — Anthrax

STUDY DESIGN:
Intervention Model Description: 3 parallel groups defined by dosing position and number of doses
Who Masked: Participant, Investigator
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- NasoShield One Dose in Position 1 (Experimental): NasoShield (1 x 10^11 vp) on Day 1 and saline placebo on Day 29 in position 1 (Group 1) in normal sitting position (no dose holding time)
  Interventions: Biological: NasoShield; Other: Placebo
- Placebo in Position 1 (Placebo Comparator): Saline placebo on Day 1 and saline placebo on Day 29 in position 1 (Group 1)
  Interventions: Other: Placebo
- NasoShield Two Doses in Position 2 (Experimental): NasoShield (1 x 10^11 vp) on Day 1 and Day 29 in position 2 (Group 2) in sitting position with nostrils elevated above head for 3 minutes followed by sitting for 27 minutes
  Interventions: Biological: NasoShield
- Placebo in Position 2 (Placebo Comparator): Saline placebo on Day 1 and Day 29 in position 2 (Group 2)
  Interventions: Other: Placebo
- NasoShield Two Doses in Position 3 (Experimental): NasoShield (1 x 10^11 vp) on Day 1 and Day 29 in position 3 (Group 3) in supine position for 30 minutes
  Interventions: Biological: NasoShield
- Placebo in Position 3 (Placebo Comparator): Saline placebo on Day 1 and Day 29 in position 3 (Group 3)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: NasoShield — NasoShield is an adenovirus-vectored anthrax vaccine
  Arms: NasoShield One Dose in Position 1; NasoShield Two Doses in Position 2; NasoShield Two Doses in Position 3
Other: Placebo — Normal saline
  Arms: NasoShield One Dose in Position 1; Placebo in Position 1; Placebo in Position 2; Placebo in Position 3

SUMMARY:
The purpose of this study is to evaluate the safety for up to two doses of NasoShield, to determine if antibodies that protect against anthrax are formed after treatment with NasoShield, and to determine whether the formation of these antibodies are affected by different positions of administration.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all healthy volunteers that have given written informed consent will undergo screening to determine eligibility for study entry. If the healthy volunteer qualifies for the study, they will be randomly assigned to 1 of 3 treatment groups. Within the treatment group, the participant will be randomized in a double-blind manner in a 5:2 ratio to NasoShield or placebo.

The investigational drug (either NasoShield or placebo) will be administered on Days 1 and 29 after qualifying into the study. The position of administration and the amount of time the subject will need to stay in the specified position will depend on the group to which the subject is assigned.

Participants will return to the investigational site for multiple visits through Day 210 (approximately 6 months after the second dose). At each visit, the participant will be asked about interim medical history and use of any medications, and safety and immunogenicity assessments will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women 18 to 49 years of age, inclusive
2. Good general health status
3. Adequate venous access for repeated phlebotomies
4. Screening laboratory results within institutional normal range or Grade 1 abnormality if the Investigator documents clinical insignificance. Creatine kinase or bilirubin may be Grade 2 if associated with normal alanine aminotransferase (ALT) and aspartate aminotransferase (AST) and the Investigator considers the result not to be clinically significant due to vigorous exercise or Gilbert's syndrome
5. Negative drug and alcohol screen at Screening and predose on Day 1
6. For women who have not been surgically sterilized or who do not have laboratory confirmation of postmenopausal status, negative pregnancy test
7. Willingness to practice a highly effective method of contraception that may include, but is not limited to, abstinence, sex only with persons of the same sex, monogamous relationship with a postmenopausal partner, monogamous relationship with vasectomized partner, vasectomy, surgical sterilization (hysterectomy, bilateral tubal ligation, salpingectomy, or oophorectomy), licensed hormonal methods, intrauterine device (IUD), or consistent use of a barrier method (eg, condom, diaphragm) with spermicide for 28 days after the last IP dose
8. Willingness to participate and comply with all aspects of the study through the entire study period, including nasopharyngeal swabs and blood and urine samples
9. Provision of written informed consent

Exclusion Criteria:

1. Pregnant, possibly pregnant, or lactating women
2. Body mass index > 35.0 kg/m2
3. Positive result for HIV, hepatitis B virus, or hepatitis C virus at Screening
4. Asthma or other chronic lung disease that is greater than mild in severity. Specifically excluded are participants with any of the following events in the past year:

   * Daily symptoms
   * Daily use of short acting beta 2 agonists
   * Use of inhaled steroids or theophylline
   * Use of pulse systemic steroids
   * Emergency care or hospitalization related to asthma or other chronic lung disease
   * Systemic steroids for asthma exacerbation
5. History of diabetes mellitus (gestational diabetes is allowed if treatment was not required postpartum and serum glucose is currently in the normal range)
6. History of coronary artery disease, arrhythmia, or congestive heart failure
7. Clinically significant ECG abnormality
8. Poorly controlled hypertension (systolic blood pressure > 150 mmHg or diastolic blood pressure > 95 mmHg) at Screening or predose on Day 1
9. History of anaphylaxis or angioedema
10. Known allergy to any of the ingredients in the vaccine formulation
11. Known allergy or sensitivity to latex
12. History of chronic rhinitis, nasal septal defect, cleft palate, nasal polyps, or other nasal abnormality that might affect vaccine administration
13. Previous nasal surgery or nasal cauterization
14. Any symptoms of upper respiratory infection or temperature > 38°C within 3 days before Day 1
15. Any symptoms within 24 hours before Day 1 of upper respiratory illness or allergy flare-up that, in the opinion of the Investigator, presents as nasal congestion or rhinorrhea that could inhibit the proper administration of the IP
16. Known or suspected malignancy, excluding non-melanoma skin cancers and other early stage surgically excised malignancies that the Investigator considers to be exceedingly unlikely to recur
17. Immunocompromised individuals, including those who have used corticosteroids(including intranasal steroids), alkylating drugs, antimetabolites, radiation, immune-modulating biologics, or other immunomodulating therapies within 90 days before Day 1 or those who plan use during the study period
18. History of autoimmune or demyelinating disease
19. Use of statin medication within 30 days before Day 1 (see list in Section 6.7.1)
20. Receipt of intranasal medications (including over-the-counter medications) within 30 days before Day 1
21. Receipt of any IP within 30 days before Day 1
22. Receipt of any vaccine within 30 days before Day 1
23. Receipt of intranasal vaccine within 90 days before Day 1
24. Receipt of any licensed or investigational anthrax vaccine in civilian or military life
25. Any change in medication for a chronic medical condition within 30 days before Day 1
26. Past regular use or current use of intranasal illicit drugs
27. Any medical, psychiatric, or social condition or occupational or other responsibility that in the judgment of the Investigator would interfere with or serve as a contraindication to protocol adherence, assessment of safety (including reactogenicity), or a subject's ability to give informed consent

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Reactogenicity to evaluate the safety of NasoShield | For 7 days after vaccination
  Subjects will record solicited local and systemic events for 7 days after each dose
Adverse Events (AEs) to evaluate the safety of NasoShield | From Day 1 to Day 210
  All adverse events from Day 1 to Day 57; serious adverse events (SAE), medically attended adverse events (MAAE), and new-onset chronic illnesses (NCI) from Day 1 to Day 210

SECONDARY OUTCOMES:
Anti-protective antigen (PA) immunoglobulin G (IgG) to evaluate humoral immunogenicity | From Day 1 to Day 210
  Titer measured by enzyme-linked immunosorbent assay (ELISA) in serum
Toxin neutralization antibody 50% neutralization factor (TNA-NF50) titer measured in serum by cytotoxic assay to evaluate humoral immunogenicity | From Day 1 to Day 210
Anti-protective antigen (PA) immunoglobulin A (IgA) to evaluate mucosal immune response | From Day 1 to Day 57
  Titer measured by enzyme-linked immunosorbent assay (ELISA) in serum

CONTACTS AND LOCATIONS:
Locations (1):
- JBR Clinical Research, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No